CLINICAL TRIAL: NCT07153263
Title: Comparison of Local Anaesthetic Spread Between the Retro-superior Costotransverse Ligament Space Block and Thoracic Paravertebral Block: A Three-dimensional CT Reconstruction Imaging Study
Brief Title: Local Anaesthetic Spread and Sensory Block Range of the Retro-superior Costotransverse Ligament Space Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Tao Shan, Attending physician, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KY 20250819-10
Record Dates: First submitted 2025-08-21; First posted 2025-09-03 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Nodules; Nerve Block
Keywords: nerve block; TPVB; ITPB; rSCTL
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- retro-SCTLB group (Experimental): A total of 20 ml of the local anesthetic solution (0.375% ropivacaine 10ml+ iohexol 10ml) is injected in the retro-superior costotransverse ligament space in the retro-SCTLB group within 60 seconds.
  Interventions: Procedure: Ultrasound-guided retro-SCTLB
- TPVB group (Experimental): A total of 20 ml of the local anesthetic solution (0.375% ropivacaine 10ml+ iohexol 10ml) is injected in the paravertebral space in the TPVB group within 60 seconds.
  Interventions: Procedure: Ultrasound-guided TPVB

INTERVENTIONS:
Procedure: Ultrasound-guided retro-SCTLB — Patients undergoing CT-guided lung nodule localization were selected for the study. Before the surgery, the retro-SCTLB was performed under ultrasound guidance.
  Arms: retro-SCTLB group
Procedure: Ultrasound-guided TPVB — Patients undergoing CT-guided lung nodule localization were selected for the study. Before the surgery, the TPVB was performed under ultrasound guidance.
  Arms: TPVB group

SUMMARY:
The aim of this clinical trial is to investigate the effects of local anesthetic diffusion range and sensory block range during retro-SCTLB(retro superior costotransverse ligament space block) and TPVB(thoracic paravertebral block) in patients undergoing CT-guided lung nodule localization. The main issue of the study is to determine the differences in the diffusion range and sensory block range of local anesthetics between the retro-SCTLB and TPVB nerve block methods.

DETAILED DESCRIPTION:
Forty patients were selected to undergo CT guided puncture localization of lung nodules under local anesthesia, and the patients were divided into groups using a computer-generated random number in a ratio of 1:1. To ensure objectivity, a nurse who was not involved in the study prepared a sealed opaque envelope containing grouping information. Patients were randomly divided into two groups: the retro-SCTLB group (group R, 20 patients), and the TPVB group (group T, 20 patients). All patients underwent ultrasound guided retro-SCTLB or TPVB before CT-guided nodule localization. Ultrasound-guided retro-SCTLB method: Using an ultrasound low-frequency convex array probe (1-6 MHZ, Sonosite, USA), the probe was placed parallel to the spine 2-3cm outside the spinous process of the fifth thoracic vertebra, on the surface of the transverse process tip. First, the probe was placed above the rib and costo-transverse process joint and observed from the inside out to clearly show the spinous process, lamina, transverse process and rib. Then, the probe was gently moved towards the caudal side. Until the sound shadows of the ribs and transverse processes disappear and inferior articular processes appear on the medial side, and when high-echo superior ligaments of the costal transverse processes appear behind the paravertebral space and anterolateral of the inferior articular processes, then gently rotate the outer edge of the probe towards the caudal side and a low-echo area can be seen behind the superior ligaments of the costal transverse processes, which is the target area. Then, using a long oblique plane puncture needle, with the in-plane technique, insert the needle from the outer side of the probe. When the needle tip reaches the target area, use the water separation technique to inject 1ml of normal saline to confirm the needle tip position, then inject 20ml of local anesthetic solution (0.375% ropivacaine 10ml+ iohexol 10ml) within 1 minute; Ultrasound-guided TPVB: Using an ultrasound low-frequency convex array probe (1-6 MHZ, Sonosite, USA), the probe is placed perpendicularly to the spine at the fifth thoracic vertebra on the midline of the trunk. First, the spinous process is identified, and then the ultrasound probe is gradually moved towards the surgical side. Structures such as the transverse process, pleura, and intercostal intima are visible. At this point, the ultrasound probe is moved parallel to the caudal side. The area between the parietal pleura, intercostal endometrium and transverse process is the target area for injection. Then, using a short inclined plane puncture needle, using the in-plane technique, the needle is inserted from the outside of the probe. When the needle tip reaches the target position, 1ml of normal saline is injected using the water separation technique to confirm the needle tip position. Then 20ml of local anesthetic solution (0.375% ropivacaine 10ml+ iohexol 10ml) is injected, and the injection is completed in 1 minute. 15 minutes after the block was completed, CT scans were performed and punctures were located, followed by three-dimensional reconstruction. Observe and record the local anesthetic solution: 1. The range of diffusion to the cranial and caudal side; 2 The range of diffusion to the intercostal space 3; The range of diffusion to the paravertebral space; 4. The range of diffusion to the epidural space; 5. The range of diffusion to the intervertebral foramen; 6. The range of diffusion to the anterolateral vertebrae (sympathetic ganglion).

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for CT-guided lung nodule localization under local anesthesia will be selected

1. aged 18-80 years
2. BMI 18-30 kg/m²
3. ASA classification I-III

Exclusion Criteria:

1. Allergy to the study drug or local anesthetic;
2. History of opioid abuse;
3. Pre-existing skin infection at the puncture site of ITPN or TPVB;
4. Peripheral infectious neuropathy;
5. Dysfunction of blood coagulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Spread of local anesthetic into the paravertebral space | 15 minutes after completion of the nerve block
  Observation of incidence and thoracic level of local anesthetic spread into the paravertebral space with CT by a researcher who was blinded to group allocation

SECONDARY OUTCOMES:
The range of the local anesthetic spreads to the intercostal space | 15 minutes after completion of the nerve block
  Observation of incidence and thoracic level of local anesthetic spread into the intercostal space with CT by a researcher who was blinded to group allocation
Observation of local anesthetic spread cephalocaudally in the erector spinae plane | 15 minutes after completion of the nerve block
  Observation of incidence and thoracic level of local anesthetic spread into the erector spinae plane cephalocaudally with CT by a researcher who was blinded to group allocation.
The range of the local anesthetic spread to the epidural space | 15 minutes after completion of the nerve block
  Observation of incidence and thoracic level of local anesthetic spread into the epidural space with CT by a researcher who was blinded to group allocation
The range of the local anesthetic spread to the anterolateral vertebrae (sympathetic ganglion). | 15 minutes after completion of the nerve block
  Observation of incidence and thoracic level of local anesthetic spread into the anterolateral vertebrae (sympathetic ganglion) with CT by a researcher who was blinded to group allocation
Assessment of skin sensory block with ice | 15 minutes after completion of the nerve block
  The sensation of skin to cold was assessed with ice. The area includes the anterior chest wall (midclavicular line), lateral chest wall (posterior axillary line), and posterior chest wall. The sensation was graded as 0 (no sensation), 1 (decreased sensation), or 2 (normal). A sensory block of the dermatome was considered to be achieved if the grade was either 0 or 1.
The range of the local anesthetic spread to the intervertebral foramen | 15 minutes after completion of the nerve block
  Observation of incidence and thoracic level of local anesthetic spread into the intervertebral foramen with CT by a researcher who was blinded to group allocation

CONTACTS AND LOCATIONS:
Overall Officials: Tao Shan, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (2):
- China (2):
  - Tao Shan, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing

IPD SHARING:
Plan to Share IPD: No